CLINICAL TRIAL: NCT04892251
Title: Ketamine Assisted Psychotherapy for Opioid Use Disorder
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00130630
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MORE+KAP (Experimental): 8 weeks of Mindfulness-Oriented Recovery Enhancement plus two ketamine assisted psychotherapy sessions
  Interventions: Combination Product: MORE+KAP
- MORE (Active Comparator): 8 weeks of Mindfulness-Oriented Recovery Enhancement
  Interventions: Behavioral: MORE

INTERVENTIONS:
Combination Product: MORE+KAP — Mindfulness-Oriented Recovery Enhancement plus two sessions where 0.5 to 1.5 mg/kg of ketamine are administered intramuscularly
  Arms: MORE+KAP
Behavioral: MORE — Mindfulness-Oriented Recovery Enhancement
  Arms: MORE

SUMMARY:
This pilot clinical trial aims to assess the preliminary efficacy of ketamine as an adjunct for a mindfulness-based intervention for opioid use disorder.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a Stage 1 randomized controlled trial to test a potential optimization of the evidence-based Mindfulness-Oriented Recovery Enhancement (MORE) intervention for opioid use disorder (OUD). Here we will add Ketamine to MORE (MORE+KAP) and test the MORE+KAP intervention versus the standard MORE intervention in a sample of patients receiving medications for OUD (MOUD; e.g, buprenorphine). The primary aim to is evaluate the extent to which MORE+KAP improves OUD treatment relative to MORE. The secondary aim is to identify the psychobiological mediators of MORE+KAP.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Opioid Use Disorder
2. Receiving OUD treatment with a buprenorphine formulation

Exclusion Criteria:

1. Previous experience with a mindfulness-based intervention program
2. Pregnancy
3. Any serious medical, mental, or cognitive issue that prevents successful participation in a mindfulness-based group treatment program
4. Prior use of ketamine other than as prescribed by a physician
5. Any of the following medical conditions

Blood Vessel Disease Heart Valve Disease Heart Failure Class 2 or Above Heart Disease Pregnancy/Breastfeeding Arteriovenous Malformation History of Intracranial Bleeding or Stroke History of Seizures Hypoxia defined by current need for supplemental oxygen Liver Disease History of allergic reaction to Ketamine Dementia (moderate-severe) History of Psychotic Disorder, Bipolar Disorder, or Personality Disorder Dissociative Identity Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Drug use | From baseline to 3-month follow-up
  Days of drug use as measured by the Timeline Followback Procedure

SECONDARY OUTCOMES:
MOUD use | From baseline to 3-month follow-up
  Days of MOUD use as measured by the Timeline Followback Procedure
Emotional Distress | From baseline to 3-month follow-up
  Emotional distress measured by the Depression Anxiety Stress Scale, range from 0 to 63, higher scores indicating worse distress.
Meaning in life | From baseline to 3-month follow-up
  Meaning in life measured by the Meaning in Life Questionnaire, Presence Subscale, range from 5 to 35, higher scores indicating more meaning in life.
Opioid craving | From baseline to 3-month follow-up
  Craving measured by the Desires for Drug Questionnaire, range from 13 to 91, higher scores indicating higher craving.
Self-transcendence | From baseline to 3-month follow-up
  Self-transcendence measured by the Nondual Awareness Dimensional Assessment, range from 13 to 65, higher scores indicating greater self-transcendence.
Affect | From baseline to 1-month follow-up
  Affect measured by Ecological Momentary Assessment, range from 0-10, higher scores indicating more intense affective states.
Mindfulness | From baseline to 3-month follow-up
  Mindfulness measured by the Five Facet Mindfulness Questionnaire, range from 39 to 195, higher scores indicating greater mindfulness.
Reappraisal | From baseline to 3-month follow-up
  Reappraisal measured by the Cognitive Emotion Regulation Questionnaire, range from 4 to 20, higher scores indicating more frequent use of reappraisal.
Savoring | From baseline to 3-month follow-up
  Savoring measured by the Brief Savoring Inventory, range from 4 to 20, higher scores indicating more use of savoring.
Momentary craving | From baseline to 1-month follow-up
  Affect measured by Ecological Momentary Assessment, range from 0-10, higher scores indicating more intense momentary craving.

OTHER OUTCOMES:
Drug cue-reactivity | From baseline to immediately after the 8 week intervention.
  Change from baseline in neurophysiological response during lab-based task involving presentation of drug cues designed to measure cue-reactivity.
Emotion regulation | From baseline to immediately after the 8 week intervention.
  Change from baseline in neurophysiological response during lab-based task involving presentation of emotional stimuli.
Theta oscillations | From baseline to immediately after the 8 week intervention.
  Theta oscillations as measured by EEG during meditation

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Garland, Principal Investigator — University of Utah
Locations (1):
- Center on Mindfulness and Integrative Health Intervention Development, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No